CLINICAL TRIAL: NCT03897374
Title: Strategic Targeting for Optimal Prevention of Cancer
Acronym: STOP-Cancer
Status: Recruiting | Type: Observational
Sponsor: ClinLogic LLC (Industry)
Collaborators: MDGlobal (Unknown)
Responsible Party: Sponsor
Other Study IDs: 02252019
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Early Detection of Cancer
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Genetic Testing — Buccal swab

SUMMARY:
The primary goal of the study is to record data over the observation period to evaluate the clinical benefit of using hereditary cancer genomic diagnostics to assess overall hereditary genetic cancer risk profile and to help guide physicians to pursue preventative measures, which may lead to early detection and treatment of the condition.

DETAILED DESCRIPTION:
Data collection will be limited to study subjects 65 years or older. The genes evaluated may be modified from time to time by the Sponsor as the body of knowledge expands and important additional pathways are identified. The list of appropriate genes that may be considered by the treating physician includes but are not necessarily limited to the following genes: ATM, BARD1, BRCA1, BRCA2, BRIP1, CDH1, CHEK2, EPCAM, MLH1, MRE11A, MSH2, MSH6, NBN, PALB2, PMS2, PTEN, RAD50, RAD51C, RAD51D, RINT1, TP53 and XRCC2. These subjects must also meet medical necessity for hereditary cancer genomic testing; and allow physician to test based on medical necessity. Hereditary Cancer testing will be diagnostic rather than screening in nature.

Study subject data will be collected only if medical necessity was established, subject agreed to test based on medical necessity and hereditary cancer genomic test was ordered by a physician related to individual study subject care considerations. The hereditary Cancer testing is independent of this data-collection, non- interventional study. The hereditary cancer genomic test must be ordered according to the individual study subject care considerations, it is not protocol specified, and will not be considered as "research" that is part of the study. Rather, the use of hereditary cancer genomic testing serves as criteria for eligibility in the study and must have been ordered for medical necessity and results received no less than 90 days prior before data is collected.

The primary goal of the study is to record data over the observation period to evaluate the clinical benefit of using hereditary cancer genomic diagnostics to assess overall hereditary genetic cancer risk profile and to help guide physicians to pursue preventative measures, which may lead to early detection and treatment of the condition; and to record physician recommended treatments and subject's brief medical history, demographic data; and investigator specialty.

Such genetic test results and recommended treatments can be tabulated and analyzed to demonstrate the clinical utility of using hereditary cancer genomic diagnostics for prevention, early detection and treatment of the condition.

The data will be collected retrospectively for a total of 120 no more than 150 days over the observation period in one (1) Case Report Form (survey). Similarly, the secondary objectives will be tabulated over the same observation period.

An interim analysis of data will be performed to determine if the study subject data collection should be increased or decreased in order to fulfill study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects may be included in the Clinical Trial if they meet all of the following inclusion criteria:

  * individuals, ages 65 years or older;
  * must have met medical necessity for hereditary cancer genomic testing and allowed the physician to test based on medical necessity;
  * hereditary cancer diagnostic test was ordered by a physician related to individual subject care considerations.
  * study subject has or had cancer
  * study subject has at least one family member with cirrent or past cancer

Exclusion Criteria:

* Study subjects will be excluded from the study if any of the following criteria apply: • study subject is currently hospitalized or incarcerated;

  * study subject is unable to provide an accurate history due to mental incapacity
  * study subject is currently abusing illicit and/or prescription drugs;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals, ages 65 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Genomic cancer screen | 120 Days
  A study subject is known to have personal and/or family history of cancer known to be influenced by genetic variation.
Genomic cancer screen | 120 Days
  A genotype known to be a predisposition for cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunbeam Clinical, Prosper, Texas, United States

IPD SHARING:
Plan to Share IPD: No